CLINICAL TRIAL: NCT06972875
Title: Efficacy and Safety of Fezolinetant for Treatment of Moderate to Severe Vasomotor Symptoms Associated With Androgen-Deprivation Therapy in Men With Prostate Cancer (FLASH): A Phase 2 Study
Brief Title: Fezolinetant for Treating Hot Flashes in Men With Prostate Cancer
Acronym: FLASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Steven Ades, Medical Oncologist, Professor of Medicine, Medical Director, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVMCC2408
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate CA; Androgen Deprivation Therapy
Keywords: prostate cancer; androgen deprivation therapy; hot flash; fezolinetant
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- fezolinetant treatment (Experimental): Adult male patients with prostate cancer experiencing hot flashes due to androgen deprivation therapy will be treated with fezolinetant. Hot flashes will be monitored to assess improvements resulting from the investigational drug
  Interventions: Drug: Fezolinetant

INTERVENTIONS:
Drug: Fezolinetant — Participants will receive fezolinetant for 28 days at FDA approved dosing and schedule of 45 mg po (per os/by mouth) once daily for treatment of hot flashes in menopausal women.

SUMMARY:
This study is for men with prostate cancer who are experiencing hot flashes due to treatments that lower testosterone. Hot flashes can affect your quality of life and make it harder for patients to continue their treatment, so researchers want to find a better way to manage them. The study is testing a drug called fezolinetant, which might help reduce hot flashes without using hormones. Fezolinetant is a drug that is currently approved for the treatment of hot flashes in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Men who are currently receiving Androgen Deprivation Therapy (ADT) for the treatment of prostate cancer. ADT is defined by a history of orchiectomy, or ongoing usage of gonadotropin-releasing hormone agonists or antagonists (e.g. leuprolide, degarelix, relugolix). Men receiving Androgen Receptor Pathway Inhibitors (ARPI) such as abiraterone, enzalutamide, apalutamide, and darolutamide are eligible.

Patients must be on a stable dose of all hormonal therapies for at least 28 days prior to registration and must not be planning to discontinue this therapy for at least 42 days following registration. Additional ARPI agents (e.g. abiraterone or enzalutamide) are allowed to be added during the Extension Phase of the trial, but not during the Treatment Phase.

Patients receiving radiation therapy during the study period are eligible. An eligible patient must have bothersome hot flashes for ≥ 7 days prior to consent, resulting in an average of four or more hot flashes per day of sufficient severity to cause the patient to seek therapeutic intervention.

Life Expectancy of 6 months or greater. Language: In order to complete the mandatory participant-completed measures, participants must be able to speak and read English.

Exclusion Criteria:

Current or future planned use of any of the following agents during the study period: drugs that are not FDA approved for use in humans, any drug with category X interactions with fezolinetant; androgens, estrogens, progesterone analogs, or complementary/alternative medicine taken for the purpose of managing hot flashes. Prior use of these agents is permitted as long as they are discontinued before registration. Stable dosing (≥ 1 month) of gabapentin, cholinergic agonists, cholinesterase inhibitors for other indications is permitted.

History of cirrhosis Elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2 X ULN or total bilirubin > ULN eGFR <30 mL/min/1.73 m2 based on reported MDRD estimate. Current use of CYP1A2 inhibitors (fezolinetant is a substrate of CYP1A2).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hot Flash Score | 28 day
  Assess the effect of fezolinetant 45 mg daily on the 7-day period participant-reported Hot Flash Score (HFS) at 4 weeks relative to baseline. The HFS sums the number of hot flashes multiplied by the intensity of each hot flash to estimate the overall hot flash burden during a 24 hour period, averaged over a 7 day period.

SECONDARY OUTCOMES:
To characterize the safety and adverse event profile of fezolinetant in the study population. | 28 day
  To characterize the safety and adverse event profile of fezolinetant in the study population by monitoring adverse events.
Measure Compliance of Fezolinetant Therapy in Men | 28 day
  Compliance will be assessed based on a combination of the Hot Flash diary (HFD) responses, the weekly phone calls during the Treatment Phase, and the participant visit at the end of the Treatment Phase.
Hot Flash Frequency | 28 day
  To assess the effect of fezolinetant on participant-reported Hot Flash Frequency (HFF) at 4 weeks relative to baseline.
Patient Reported Quality of Life | 28 day
  To measure the impact of fezolinetant treatment participant-reported quality of life and hot flash interference, as measured by the Hot Flash Related Daily Interference Scale (HFRDIS) after 4 weeks compared to baseline. The HFRDIS is a 10-item instrument developed and validated to assess the interference of hot flashes on multiple specific important quality of life dimensions in this patient population.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No